CLINICAL TRIAL: NCT05643599
Title: The Relationship Between Oxidative Stress and Apoptosis of Histopathological Changes Made by Mad Honey Containing Grayanotoxin in the Ovary
Brief Title: The Relationship With Mad Honey Containing Grayanotoxin and Ovary Tissue
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Hayrunnisa Yesil Sarsmaz, Asistant Prof., Celal Bayar University
Other Study IDs: MCBU_Madhoney
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Ovary Disease
Keywords: Grayonotoxin; Mad Honey; Normal honey; ovary
MeSH Terms: conditions — Ovarian Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ovary tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1:: Mad honey
  Interventions: Dietary Supplement: Mad Honey
- Group 2:: Normal honey
  Interventions: Dietary Supplement: Normal Honey
- Group 3:: without intervention
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Mad Honey — mad honey (80 mg/kg); (n:6)
  Groups: Group 1:
Dietary Supplement: Normal Honey — normal honey (80 mg/kg),(n:6)
  Groups: Group 2:
Dietary Supplement: Control — Control
  Groups: Group 3:

SUMMARY:
For our working group, eighteen healthy Sprague-Dawley female rats were recruited and separated into three groups in an experimental animal laboratory.

Group 1 was given mad honey (n:6) (80 mg/kg); Group 2 was given normal honey (n:6) (80 mg/kg), and Group 3 was the control group (n:6). The groups were given normal and mad honey by oral gavage for 30 days in this study. Rats were anesthetized intramuscularly with 50 mg/kg ketamine and 5 mg/kg xylazine on the 30th day of the study. At the conclusion of the study, female rats in the proestrus phase of the estrous cycle (as indicated by vaginal smear) were sacrificed and their ovarian tissues were placed in neutral formalin solution.

DETAILED DESCRIPTION:
Honey poisoning is caused by consuming honey produced by bees that feed on Rhododendron family plants. Rhododendron poisoning goes by names such as mad honey poisoning or grayanotoxin poisoning. The purpose of this study is to determine the effects of grayanotoxin in mad honey on ovarian tissue folliculogenesis in terms of cell death and nitric oxide expression. Three groups of 18 female Sprague-Dawley rats were formed. The first group received mad honey (80 mg/kg), the second group received normal honey (80 mg/kg), and the third group is control. The first and second groups received normal and mad honey by oral gavage for 30 days before being sacrificed under anesthesia The caspase 3 immunostaining group observed a moderate to a strong response, particularly in the granulosa cells of the Graaf follicles in the mad honey group, while the normal honey and control groups observed a weak to moderate reaction. In the mad honey group, immunostaining for caspase8 and caspase 9 revealed a moderate immunoreaction in the granulosa cells of the Graaf follicles, while expression was weak in the normal honey and control groups. The TUNEL approach revealed that the majority of Graaf follicles that exhibited TUNEL positive in the mad honey group and progressed to atresia were Graaf follicles. The iNOS immunoreaction revealed a high level of expression in the mad honey group, particularly in several Graaf follicles. In all three groups, a weak reactivity to eNOS immunostaining was seen in both Graaf follicles and theca external layers. According to the findings of apoptotic and nitric oxide marker expression, it was determined that mad honey may result in an increase in follicular atresia in ovarian follicles when compared to normal honey and control groups.

ELIGIBILITY:
Inclusion Criteria:

* healthy rats

Exclusion Criteria:

* patient rats
* not eating rats

Ages: 8 Weeks to 10 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: experimental animals ( Sprague Dawley rats)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the Mad Honey and Normal Honey findings of the ovary tissue specimens | Baseline
  Analyses of the relationship between oxidative stress and apoptosis of histopathological changes made by mad honey containing grayanotoxin in the ovary

CONTACTS AND LOCATIONS:
Overall Officials: Gulsen Gurgen, Study Chair — Manisa Celal Bayar University; Suha Turkmen, Study Chair — Karadeniz Teknik University
Locations (1):
- Hayrunnisa, Yunusemre, Mani̇sa, Turkey (Türkiye)